CLINICAL TRIAL: NCT05221619
Title: Nipocalimab Post-trial Access in Patients With Warm Autoimmune Hemolytic Anemia (wAIHA) Who Are Experiencing Clinical Benefit After Complete 28-Weeks Open-label Extension in MOM-M281-006
Brief Title: Post-trial Access for Nipocalimab in Participants With Warm Autoimmune Hemolytic Anemia (wAIHA)
Status: Temporarily not available | Type: Expanded Access
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR109152; 80202135WHA4001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2022-01-05; First posted 2022-02-03 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Warm Autoimmune Hemolytic Anemia

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Nipocalimab — Depending on the dose received at their last administration in the MOM-M281-006 (NCT04119050) study, participants will continue to receive either nipocalimab dose-1 every 2 weeks (Q2W) or nipocalimab dose-2 every 4 weeks (Q4W) by intravenous (IV) infusion.
  Other Names: M281; JNJ-80202135

SUMMARY:
The purpose of this post-trial access (PTA) program is to provide nipocalimab for the treatment of participants with Warm Autoimmune Hemolytic Anemia (wAIHA) who are experiencing clinical benefit after completing 28-weeks open-label extension in MOM-M281-006 (NCT04119050) study.

ELIGIBILITY:
Inclusion Criteria:

* Participants demonstrate clinical benefit (improvement of hemoglobin from baseline) at the Week 28 assessment in the open-label extension of the MOM-M281-006 (NCT04119050) study
* Participants does not have co-morbidities that would alter the risk-benefit of nipocalimab administration (determined by treating physician)
* Participants completed treatment in the 28-week open-label extension of the MOM-M281-006 (NCT04119050) study without receiving rescue treatment or discontinuation of the study prior to Week 28 visit

Exclusion Criteria:

* Participants have a serious or clinically significant infection (example: pneumonia, biliary tract infection, diverticulitis, Clostridioides difficile infection) requiring parenteral anti-infectives and/or hospitalization
* Participants have a chronic infection (example: bronchiectasis, chronic osteomyelitis, chronic pyelonephritis) or require chronic treatment with anti-infectives (example: antibiotics, antivirals)

Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC